CLINICAL TRIAL: NCT06440317
Title: Investigation of Immunothrombosis in Intensive Care Patients With Septic Shock Undergoing Renal Replacement Therapy With the OXIRIS Membrane
Brief Title: Immunothrombosis With Septic Shock Undergoing Renal Replacement Therapy With the OXIRIS Membrane
Acronym: PLAQSIRIS
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Bordeaux (Other)
Collaborators: Baxter Healthcare Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: CHUBX 2023/93
Record Dates: First submitted 2024-04-25; First posted 2024-06-03 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Sepsis
Keywords: Intensive Care; Immunothrombosis; NETs; Neutrophils; Platelets
MeSH Terms: conditions — Sepsis; Thromboinflammation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples will be collected in citrate and EDTA tubes before and after the membrane on the day of initiating renal replacement therapy (Day 0), the day after starting therapy (Day 1), and 5 days after (Day 5). Extraction of peripheral blood mononuclear cells (PBMCs) will be done.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Hemofiltration membranes (the oXiris® membrane and the HF1400 ® membrane): Eligible patients for this study will undergo renal replacement therapy using two hemofiltration membranes commonly used in intensive care units.
  Interventions: Device: Hemofiltration membranes (the oXiris membrane® and the HF1400® membrane)

INTERVENTIONS:
Device: Hemofiltration membranes (the oXiris membrane® and the HF1400® membrane) — The PRISMAFLEX® or PRISMAX® control unit (pre- and post-dilution with a prescribed treatment dose > 25 ml/kg/h) with regional citrate anticoagulation and a substitution solution by PHOXILLUM will be used regardless of the type of membrane used (the oXiris membrane and the HF 1400 membrane), also as part of routine care provided in the ICU.

SUMMARY:
Sepsis remains a global scourge. Before the SARS-CoV-2 pandemic, the World Health Organization estimated approximately 49 million cases annually, resulting in 11 million deaths. Defined by dysregulated host response to infection, sepsis leads to vital organ failure. Renal dysfunction affects about half of ICU patients, necessitating extracorporeal renal replacement therapy in approximately 10% of cases, alongside coagulation system involvement typified by thrombocytopenia. Immunothrombotic phenomena are pivotal in sepsis pathophysiology, activating coagulation and disrupting immune responses. Microcirculatory impairment, mediated by neutrophils, monocytes, and platelets, worsens vital organ perfusion. Excessive production of Neutrophil Extracellular Traps (NETs) is implicated in microcirculatory compromise during sepsis.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years and older
* Admitted to the intensive care unit with septic shock, defined as an increase in the Sequential Organ Failure Assessment (SOFA) score of at least 2 points due to infection, requiring vasopressor drugs to maintain a mean arterial pressure (MAP) ≥ 65 mmHg, and a lactate level > 2 mmol/L (18 mg/dL) despite adequate fluid resuscitation
* Requiring renal replacement therapy according to consensus indications:

  * KDIGO stage 3 acute kidney injury with oliguria or anuria persisting for more than 72 hours
  * Urea > 40 mmol/L
  * Plasma potassium > 5.5 mmol/L despite medical treatment
  * pH < 7.15 (pure metabolic acidosis with PaCO2 < 30 mmHg or mixed acidosis with PaCO2 > 50 mmHg without the possibility of improving alveolar ventilation)
  * Acute pulmonary edema secondary to hydrosaline overload resulting in severe hypoxemia (oxygen flow > 5 L/min or FiO2 > 50% during mechanical ventilation to maintain SaO2 > 95%) despite diuretic therapy
* Receiving continuous renal replacement therapy with a high-adsorption membrane (oXiris membrane) or a conventional membrane (HF1400 membrane)

Exclusion Criteria:

* Known history of constitutional thrombopathy (Bernard Soulier disease, Glanzmann thrombasthenia, Gray's syndrome or dense granule disease)
* Myelodysplastic or myeloproliferative syndrome
* Autoimmune thrombocytopenic purpura
* Acute leukemia
* Hemorrhagic shock
* Platelet transfusion within 7 days prior to inclusion
* Antiplatelet therapy with clopidogrel or ticagrelor within 5 days prior to inclusion, prasugrel or dipyridamole within 7 days prior to inclusion
* Active HIV infection or hepatitis B or C
* Pregnant woman
* Not affiliated to a social security system or not benefiting from such a system

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Eligible patients for this study will undergo renal replacement therapy using two hemofiltration membranes commonly used in intensive care units
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2026-04 (Estimated); Primary Completion 2027-04 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Immunothrombosis : Concentration of platelet activation markers | 12 months after inclusion day
  Dosages of platelet activation markers, before and after the renal replacement therapy membrane : oXiris membrane or conventional membrane

SECONDARY OUTCOMES:
NETosis : Concentration of Neutrophil Extracellular Traps | 12 months after inclusion day
  Dosages of Neutrophil Extracellular Traps, before and after the renal replacement therapy membrane : oXiris membrane or conventional membrane
Monocyte activation : Concentration of monocyte (CD14+) | 12 months after inclusion day
  Dosages of monocyte (CD14+), before and after the renal replacement therapy membrane : oXiris membrane or conventional membrane

CONTACTS AND LOCATIONS:
Overall Officials: Maria MAMANI, Pr, Study Chair — ImmunoConcEpT, Bordeaux University
Locations (1):
- Hopital Haut-Lévêque, Pessac, France